CLINICAL TRIAL: NCT03549650
Title: Prevention and Management of Intravesical BCG-related Lower Urinary Tract Symptoms With Prophylactic Pentosan Polysulphate in Patients With Non-Muscle-Invasive Bladder Cancer: A Randomized Controlled Trial
Brief Title: Prevention and Management of Intravesical BCG-related Lower Urinary Tract Symptoms
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Given the updated precautions on Elmiron as well as the risk benefit profile, we have decided to terminate the study.
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Collaborators: Cancer Research Network (Other)
Responsible Party: Principal Investigator, Lysanne Campeau, MDCM, PhD, FRCSC, Assistant Professor, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17-149
Record Dates: First submitted 2018-04-23; First posted 2018-06-08 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Lower Urinary Tract Symptoms; Bladder Carcinoma; BCG
Keywords: Non-Muscle-Invasive Bladder Cancer; LUTS
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — Capsules; Pentosan Sulfuric Polyester; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pentosan Polysulfate Na 100Mg Cap (Experimental): Drug intervention of Pentosan Polysulfate Na 100Mg Cap (ELMIRON) thrice daily PO for 6 weeks, after meeting the eligibility criteria during the the two-week Screening period.
  Interventions: Drug: Pentosan Polysulfate Na 100Mg Cap
- Placebo oral capsule (Placebo Comparator): Participants will receive Placebo oral capsule, similar to (ELMIRON 100mg) thrice daily PO for 6 weeks, , after meeting the eligibility criteria during the the two-week Screening period.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Pentosan Polysulfate Na 100Mg Cap — Participants will be randomly assigned to receive Pentosan Polysulfate Na 100Mg Cap TID for 6 weeks.
  For blinded distribution, each bottle of medications will be labeled with a random number for identification.
  The study participants will be monitored every 2 weeks with phone calls from the study team to evaluate their condition and decide if the medication is tolerated and whether it should be continued or stopped.
  Other Names: ELMIRON
  Arms: Pentosan Polysulfate Na 100Mg Cap
Drug: Placebo oral capsule — Participants will be randomly assigned to receive Placebo oral capsule TID for 6 weeks.
  For blinded distribution, each bottle of medications will be labeled with a random number for identification.
  The study participants will be monitored every 2 weeks with phone calls from the study team to evaluate their condition and decide if the medication is tolerated and whether it should be continued or stopped.
  Other Names: Sugar pill
  Arms: Placebo oral capsule

SUMMARY:
Common local side effects are generally seen during induction and during the first 6 months of BCG maintenance. BCG-related cystitis is frequent and unavoidable. Furthermore, repeated BCG instillation increases the incidence and severity of irritative bladder symptoms. Several methods attempted to reduce the intensity and frequency of BCG- related lower urinary tract symptoms (LUTS), such as, administration of anti-tuberculosis drug isoniazid or oral antibiotic ofloxacin or by reducing the BCG dose, but without any encouraging results. Local side effects requiring cessation of treatment are seen more frequently in the first year of therapy, preventing patients from receiving their BCG maintenance regimen.

Pentosan Polysulphate (PPS), is an oral medication with unique analgesic properties used to relieve bladder pain and discomfort related to other conditions, has been investigated in a small study with encouraging result in this patient population. This suggest that PPS is well tolerated and effective at decreasing BCG-related LUTS.

The purpose of this study is first to investigate the efficacy of co-administration of Pentosan Polysulphate to prevent these adverse events and the impact of this intervention on quality of life. The second goal is to determine which patients are more vulnerable to develop BCG- related lower urinary tract symptoms (LUTS), based on clinical assessment, demographics data, voiding parameters, and urinary inflammatory markers, and then to assess the effectiveness of BCG therapy following co-administration of ELMIRON.

DETAILED DESCRIPTION:
Study purpose and rationale:

BCG-related LUTS is a condition which can have a significant negative impact on the psychological well-being, social functioning, and overall quality of life of bladder cancer patients. Clinical studies have demonstrated effects of PPS on damaged urothelium in the bladder, which is a key feature for diminishing BCG local side effects. The "dual action" protective effect on bladder epithelium and replacing the mucus in the glycosaminoglycan layer of damaged urothelium provides a scientific rationale to evaluate whether PPS treatment may be a preventive option for NMIBC patients treated with BCG.

It is therefore important to find a treatment strategy to control the BCG-related LUTS so that candidate patients do not lose the benefit of BCG treatment while maintaining its efficacy and ensuring optimal outcomes. This study will identify the patients that are more vulnerable to develop these side effects and determine the efficacy of PPS to diminish BCG- related lower urinary tract symptoms (LUTS) and associated impact on quality of life.

Sample Size:

For the first aim, power analysis was estimated using a One-way (ANOVA) hypothesis test with a type 1 error of 5%, 80% power, and 20% dropout rate. It was calculated based on the ICIQ-LUTSqol expected values. The baseline mean ICIQ-LUTSqol score used was 33.1 and SD of 7.3, the outcome ICIQ-LUTSqol score mean used 28.48, with a SD of 4.95, which is the minimally important difference of 3.7124. The investigator calculate a number of 30 patients per group, for a total sample size of 60. (Calculated by pass program v 15.0.03)

For the second aim, a total number of 40 candidates will be recruited for this prospective study. The investigator expect a minimum of 30% of patients to experience BCG related LUTS, therefore 18 patients with LUTS The SD of ICIQ-LUTSqol is 7.3 and its maximum score is 76. Therefore, the investigator estimate a required sample size of 14 (1.96 2 SD 2 / 3.82), for a p value < 0.05, and an absolute error of 0.05.

The comparison between groups of the cohort will be conducted using chi-square analysis. A 2-sample t test will be used to compare baseline scores between study groups. The Wilcoxon rank-sum test will be used to calculate whether the mean difference of all the outcome measures between groups. A p value <0.05 considered statistically significant.

Approximately 100 subjects are expected to be enrolled for this prospective trial. It is expected that 20% of subjects will not qualify for randomization after screening. The study is expected to randomize approximately 80 subjects into the double-blind treatment where subjects will be allocated to ELMIRON 100 mg, or matched placebo TID in a 1:1 ratio. A post randomisation dropout rate of 20% has been estimated, resulting in 60 evaluable subjects. This provides an 80% power for the primary endpoint.

Study design and description This is a Phase 2, double-blind, randomized, placebo-controlled, parallel-group study in patients 18 to 85 years old with NMIBC. The study will include a two weeks Screening Period; and a 6-week double-blind Treatment Period. Participants will return to the clinic for a safety Follow-up Visit 6 and 18 weeks after treatment is completed for a total study duration of 24 weeks.

All participants will enter the Screening Period during which eligibility will be assessed, where subjects must have at least 3 days of daily diary symptom collection. Participants who continue to meet eligibility criteria, including collection of diary data, Negative Urine analysis and culture, and bladder scan showing PVR less than 150ml at the end of the Screening Period will enter the Treatment Period.

Participants will be randomly assigned (1:1) to receive study drug (ELMIRON 100 mg, or placebo) TID for a duration of 6weeks.

Efficacy will be assessed by number of urgency episodes per 24 hours based on a 3-day bladder diary, the Overactive Bladder-Validated 8- Question (OAB-V8), the visual analogue scale for suprapubic and perineal pain (VAS), the ICIQ-Lower Urinary Tract Symptoms Quality of Life Questionnaire (ICIQ-LUTSqol), and quantitative measures of urinary inflammatory markers levels (TRAIL, IFN, IL-2, IL-10).

Safety assessments will be conducted throughout the trial and will include physical examinations, vital signs, clinical laboratory evaluations, cystoscopy, urine cytology, and adverse events (AEs).

Study conduct:

AIM 1: Determine the effectiveness of co-administration of Pentosan Polysulphate in preventing BCG-related LUTS.

Rationale: The investigator aim to compare the effect of PPS (ELMIRON) to placebo on the incidence and severity of local adverse effects of BCG intravesical therapy and its impact on health-related quality of life (HRQoL) in patients with superficial bladder cancer. As the currently used symptomatic treatment drugs failed to prove optimal efficacy, new treatment options are warranted. PPS could be a promising drug especially when considering its effectiveness in controlling LUTS related to similar pathologies.

The first aim will be a prospective, randomized, double-blinded, placebo-controlled pilot study, A total of 60 subjects will be assessed and included in the study after obtaining their consent and fulfilling the inclusion criteria. Within 14 days after TURBT, patients will undergo baseline evaluation and will be randomized into two groups as the following:

* Group A will receive PPS 100 mg (ELMIRON) thrice daily PO. (30 subjects)
* Group B will receive placebo thrice daily PO. (30 subjects) Treatment period for all groups will be 6 weeks as co-administration with BCG instillation.

AIM 2: Identify predisposing factors to developing BCG-related LUTS based on clinical, demographic and voiding parameters The second aim will involve an in-depth pre-treatment analysis of clinical parameters of patients planned for BCG instillation and correlation with the development of BCG local side effects. Prior to receiving BCG induction, patients will be evaluated for baseline demographics, voiding diary, non-invasive uroflowmetry with post-void residual, LUTS and quality of life questionnaires (OAB-V8, ICIQ-LUTSqol, and VAS). Objective outcomes assessment using quantitative measures of TRAIL, IFN, IL-2, and IL-10 levels in the urine before and following BCG induction treatment will be quantitated using a sandwich ELISA and correlated with the severity of LUTS. This prospective cohort will be followed 3 months after completing the induction phase by repeating the clinical assessment described and identify their oncological response to the treatment by urine cytology/cystoscopy.

Confidentiality:

All study outcomes and documents will be considered as confidential. The Investigator and members of his/her research team must not disclose such information without prior written authorization. The anonymity of participating patients must be maintained. Subjects will be identified on CRFs and other documents by their subject number/code, not by name. Documents that identify the subject (eg, the signed informed consent) must be retained in confidence by the Investigator. All data will remain confidential and will be available for access by the investigators only. A unique identifier to keep their identity confidential will identify the participant. The information will be kept for duration of 10 years.

Statement on ethical consideration:

The proposed study protocol ensures that the Sponsor and Investigator adhere to the principles of the GCP guidelines of the ICH, and of the recent version of the Declaration of Helsinki. The study also will be following with local ethics requirements.

ELIGIBILITY:
Inclusion Criteria:

Adult patients aged 18 to 85 will be eligible for inclusion in this study if all of the following criteria apply:

1. Willing to provide written informed consent
2. Confirmed diagnosis (biopsy-proven) of intermediate- and high-risk NMIBC
3. Two to four weeks following complete tumor resection
4. Candidate for BCG induction therapy based on CUA clinical guidelines
5. Subjects must not be pregnant, lactating, or actively trying to become pregnant, Subjects who are premenopausal and of childbearing potential must have a negative pregnancy test at Screening (serum) and at Day 0 (urine) and must use a medically acceptable and effective method of birth control for the duration of the study, which can include:

   1. Having a male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject
   2. Use of double-barrier methods of contraception; condoms with the use of caps (with spermicide) and intra-uterine devices are acceptable
   3. Use of hormonal contraceptives (oral, depots, patches, etc.) with double-barrier methods of contraception as outline above
   4. True abstinence: When this is in line with the preferred and usual lifestyle of the subject (period abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)

Exclusion Criteria:

1. Contraindications to BCG therapy
2. Solitary tumors except pT1 high grade
3. Tumor stage ≥ T2
4. Previous BCG or chemotherapy instillation
5. Carcinoma in situ and variant histology of urothelial carcinoma
6. Subjects with concurrent (at Screening), urinary tract infections (positive dipstick for urinary tract infection and abnormal microscopic evaluation, signs and symptoms)
7. Unevaluated urinary retention, Post void residual (PVR) urine volume > 150 ml
8. Diagnosis of dementia
9. Any concurrent condition or any clinically significant abnormality on the screening physical examination, laboratory tests, which, in the opinion of the Investigator, may affect the interpretation of efficacy or safety data, or which otherwise contraindicates participation in a clinical study with PPS.

   1. Hypersensitivity to PPS or any of its ingredients
   2. History of clinically significant drug hypersensitivity.
   3. Clinically significant or unstable, endocrine, hepatic, renal, immunologic, or heart disease
   4. Patients at increased hemorrhagic risk due to unstable disease course (ulcerative GI lesions, aneurysms, internal or external hemorrhoids, thrombocytopenia, hemophilia, polyps or diverticulae).
10. Use of any pharmacologic agent used to treat symptoms of LUTS
11. Participation in a clinical study within the month prior to screening, or exposure to an investigational drug which has not washed out since the last administration prior to screening
12. In the opinion of the Investigator, is at risk of non-compliance with study procedures, or cannot read, understand, or complete study-related materials, particularly informed consent
13. Participation in any clinical study of an investigational drug that may affect urinary function within 1 months prior to screening
14. Severe renal impairment (estimated glomerular filtration rate < 30 mL/min/1.73m2)
15. Severe hepatic impairment (Child-Pugh B or greater)
16. You are pregnant or breastfeeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy (Urgency episodes assessed by bladder diary) a of co-administration of Pentosan Polysulphate in preventing BCG-related LUTS in adult subjects with a diagnosis of NMIBC. | Start of treatment to End of treatment (6weeks)
  Primary outcome assessment (change from baseline to end of treatment):
  -Mean change in number of urgency episodes per 24 hours based on a 3-day bladder diary
Determine the efficacy (Urgency episodes assessed by ICIQ-LUTSqol questionnaire) a of co-administration of Pentosan Polysulphate in preventing BCG-related LUTS in adult subjects with a diagnosis of NMIBC. | Start of treatment to End of treatment (6weeks)
  Primary outcome assessment (change from baseline to end of treatment):
  -Mean change in ICIQ-LUTSqol questionnaire score
Determine the efficacy (Urgency episodes assessed by OAB-V8 questionnaire) a of co-administration of Pentosan Polysulphate in preventing BCG-related LUTS in adult subjects with a diagnosis of NMIBC. | Start of treatment to End of treatment (6weeks)
  Primary outcome assessment (change from baseline to end of treatment):
  -Mean change in OAB-V8 questionnaire score
Determine the safety (Adverse events or reactions as assessed by CTCAE v5.0) of co-administration of Pentosan Polysulphate in preventing BCG-related LUTS in adult subjects with a diagnosis of NMIBC. | Start of treatment to End of treatment (6weeks)
  Safety: (Number of participants with treatment-related adverse events as assessed by CTCAE v5.0)
  -Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 at the End of treatment Visit (week 6)

SECONDARY OUTCOMES:
Efficacy of BCG therapy (cancer recurrence and progression assessed by cystoscopy) following co-administration of Pentosan Polysulphate | 12 weeks and 24 weeks
  All patients will be also evaluated at 12 and 24 weeks by cystoscopy to evaluate the impact of this intervention on the efficacy of BCG therapy as well as to check for cancer recurrence and progression as routine standard of care
Efficacy of BCG therapy (cancer recurrence and progression assessed by urine cytology) following co-administration of Pentosan Polysulphate | 12 weeks and 24 weeks
  All patients will be also evaluated at 12 and 24 weeks by urine cytology to evaluate the impact of this intervention on the efficacy of BCG therapy as well as to check for cancer recurrence and progression as routine standard of care
Predisposing factors to developing BCG-related LUTS involving secondary analysis of patient's characteristics pre- and post-treatment | Start of treatment to End of treatment (6weeks)
  This will involve an in-depth pre-treatment analysis of clinical parameters of patients planned for BCG instillation and correlation with the development of BCG local side effects
Predisposing factors to developing BCG-related LUTS evaluated by ELISA quantitative measures of urinary inflammatory markers before and after BCG therapy | Start of treatment to End of treatment (6weeks)
  Objective outcomes assessment using quantitative measures of TRAIL, IFN, IL-2, and IL-10 levels in the urine before and following BCG induction treatment will be quantitated using a sandwich ELISA and correlated with the severity of LUTS
Health-related quality of life (HRQoL) assessed by ICIQ-LUTSqol questionnaire | Baseline, 6weeks , 12 weeks and 24 weeks
  Assess the impact of this intervention on Health-related quality of life (HRQoL) in bladder cancer patients using quality of life questionnaire ICIQ-LUTSqol
Health-related quality of life (HRQoL) assessed by VAS questionnaire | Baseline, 6weeks , 12 weeks and 24 weeks
  Assess the impact of this intervention on Health-related quality of life (HRQoL) in bladder cancer patients using quality of life questionnaire VAS

CONTACTS AND LOCATIONS:
Overall Officials: Lysanne Campeau, MD, PhD, Principal Investigator — SirMortimer JGH
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brausi M, Witjes JA, Lamm D, Persad R, Palou J, Colombel M, Buckley R, Soloway M, Akaza H, Bohle A. A review of current guidelines and best practice recommendations for the management of nonmuscle invasive bladder cancer by the International Bladder Cancer Group. J Urol. 2011 Dec;186(6):2158-67. doi: 10.1016/j.juro.2011.07.076. Epub 2011 Oct 19. PMID 22014799
- [Background] Gontero P, Bohle A, Malmstrom PU, O'Donnell MA, Oderda M, Sylvester R, Witjes F. The role of bacillus Calmette-Guerin in the treatment of non-muscle-invasive bladder cancer. Eur Urol. 2010 Mar;57(3):410-29. doi: 10.1016/j.eururo.2009.11.023. Epub 2009 Nov 13. PMID 19969411
- [Background] Lamm DL, van der Meijden PM, Morales A, Brosman SA, Catalona WJ, Herr HW, Soloway MS, Steg A, Debruyne FM. Incidence and treatment of complications of bacillus Calmette-Guerin intravesical therapy in superficial bladder cancer. J Urol. 1992 Mar;147(3):596-600. doi: 10.1016/s0022-5347(17)37316-0. PMID 1538436
- [Background] Brausi M, Oddens J, Sylvester R, Bono A, van de Beek C, van Andel G, Gontero P, Turkeri L, Marreaud S, Collette S, Oosterlinck W. Side effects of Bacillus Calmette-Guerin (BCG) in the treatment of intermediate- and high-risk Ta, T1 papillary carcinoma of the bladder: results of the EORTC genito-urinary cancers group randomised phase 3 study comparing one-third dose with full dose and 1 year with 3 years of maintenance BCG. Eur Urol. 2014 Jan;65(1):69-76. doi: 10.1016/j.eururo.2013.07.021. Epub 2013 Jul 24. PMID 23910233
- [Background] de Reijke TM, de Boer EC, Kurth KH, Schamhart DH. Urinary cytokines during intravesical bacillus Calmette-Guerin therapy for superficial bladder cancer: processing, stability and prognostic value. J Urol. 1996 Feb;155(2):477-82. PMID 8558640
- [Background] Ludwig AT, Moore JM, Luo Y, Chen X, Saltsgaver NA, O'Donnell MA, Griffith TS. Tumor necrosis factor-related apoptosis-inducing ligand: a novel mechanism for Bacillus Calmette-Guerin-induced antitumor activity. Cancer Res. 2004 May 15;64(10):3386-90. doi: 10.1158/0008-5472.CAN-04-0374. PMID 15150089
- [Background] Sylvester RJ, Brausi MA, Kirkels WJ, Hoeltl W, Calais Da Silva F, Powell PH, Prescott S, Kirkali Z, van de Beek C, Gorlia T, de Reijke TM; EORTC Genito-Urinary Tract Cancer Group. Long-term efficacy results of EORTC genito-urinary group randomized phase 3 study 30911 comparing intravesical instillations of epirubicin, bacillus Calmette-Guerin, and bacillus Calmette-Guerin plus isoniazid in patients with intermediate- and high-risk stage Ta T1 urothelial carcinoma of the bladder. Eur Urol. 2010 May;57(5):766-73. doi: 10.1016/j.eururo.2009.12.024. Epub 2009 Dec 18. PMID 20034729
- [Background] Vegt PD, van der Meijden AP, Sylvester R, Brausi M, Holtl W, de Balincourt C. Does isoniazid reduce side effects of intravesical bacillus Calmette-Guerin therapy in superficial bladder cancer? Interim results of European Organization for Research and Treatment of Cancer Protocol 30911. J Urol. 1997 Apr;157(4):1246-9. PMID 9120912
- [Background] Colombel M, Saint F, Chopin D, Malavaud B, Nicolas L, Rischmann P. The effect of ofloxacin on bacillus calmette-guerin induced toxicity in patients with superficial bladder cancer: results of a randomized, prospective, double-blind, placebo controlled, multicenter study. J Urol. 2006 Sep;176(3):935-9. doi: 10.1016/j.juro.2006.04.104. PMID 16890660
- [Background] Oddens J, Brausi M, Sylvester R, Bono A, van de Beek C, van Andel G, Gontero P, Hoeltl W, Turkeri L, Marreaud S, Collette S, Oosterlinck W. Final results of an EORTC-GU cancers group randomized study of maintenance bacillus Calmette-Guerin in intermediate- and high-risk Ta, T1 papillary carcinoma of the urinary bladder: one-third dose versus full dose and 1 year versus 3 years of maintenance. Eur Urol. 2013 Mar;63(3):462-72. doi: 10.1016/j.eururo.2012.10.039. Epub 2012 Nov 2. PMID 23141049
- [Background] Anderson VR, Perry CM. Pentosan polysulfate: a review of its use in the relief of bladder pain or discomfort in interstitial cystitis. Drugs. 2006;66(6):821-35. doi: 10.2165/00003495-200666060-00006. PMID 16706553
- [Background] Teichman JM. The role of pentosan polysulfate in treatment approaches for interstitial cystitis. Rev Urol. 2002;4 Suppl 1(Suppl 1):S21-7. PMID 16986030
- [Background] Yadav S, Tomar V, Yadav SS, Priyadarshi S, Banerjee I. Role of oral pentosan polysulphate in the reduction of local side effects of BCG therapy in patients with non-muscle-invasive bladder cancer: a pilot study. BJU Int. 2016 Nov;118(5):758-762. doi: 10.1111/bju.13489. Epub 2016 Apr 23. PMID 27010115
- [Background] Davis EL, El Khoudary SR, Talbott EO, Davis J, Regan LJ. Safety and efficacy of the use of intravesical and oral pentosan polysulfate sodium for interstitial cystitis: a randomized double-blind clinical trial. J Urol. 2008 Jan;179(1):177-85. doi: 10.1016/j.juro.2007.08.170. Epub 2007 Nov 14. PMID 18001798
- [Background] Chuang YC, Lee WC, Lee WC, Chiang PH. Intravesical liposome versus oral pentosan polysulfate for interstitial cystitis/painful bladder syndrome. J Urol. 2009 Oct;182(4):1393-400. doi: 10.1016/j.juro.2009.06.024. Epub 2009 Aug 15. PMID 19683290
- [Background] Grigsby PW, Pilepich MV, Parsons CL. Preliminary results of a phase I/II study of sodium pentosanpolysulfate in the treatment of chronic radiation-induced proctitis. Am J Clin Oncol. 1990 Feb;13(1):28-31. doi: 10.1097/00000421-199002000-00008. PMID 1689537
- [Background] De Reijke TM, De Boer LC, Steerenberg PA, Vos PC, Kurth KH, Schamhart DH. The effects of intravesical pretreatment with pentosan polysulfate on the bacillus Calmette-Guerin induced immune reaction of the guinea pig. J Urol. 1994 Mar;151(3):746-9. doi: 10.1016/s0022-5347(17)35079-6. PMID 7508528
- [Background] Schamhart DH, de Boer EC, Kurth KH. Interaction between bacteria and the lumenal bladder surface: modulation by pentosan polysulfate, an experimental and theoretical approach with clinical implication. World J Urol. 1994;12(1):27-37. doi: 10.1007/BF00182048. PMID 7516779
- [Background] Abdo KM, Johnson JD, Nyska A. Toxicity and carcinogenicity of Elmiron in F344/N rats and B6C3F1 mice following 2 years of gavage administration. Arch Toxicol. 2003 Dec;77(12):702-11. doi: 10.1007/s00204-003-0472-9. Epub 2003 Sep 24. PMID 14508637
- [Background] National Toxicology Program. NTP technical report on the toxicology and carcinogenesis studies of 2,3,7,8-tetrachlorodibenzo-p-dioxin (TCDD) (CAS No. 1746-01-6) in female Harlan Sprague-Dawley rats (Gavage Studies). Natl Toxicol Program Tech Rep Ser. 2006 Apr;(521):4-232. PMID 16835633
- [Background] Kassouf W, Traboulsi SL, Kulkarni GS, Breau RH, Zlotta A, Fairey A, So A, Lacombe L, Rendon R, Aprikian AG, Siemens DR, Izawa JI, Black P. CUA guidelines on the management of non-muscle invasive bladder cancer. Can Urol Assoc J. 2015 Sep-Oct;9(9-10):E690-704. doi: 10.5489/cuaj.3320. Epub 2015 Oct 13. No abstract available. PMID 26664503
- [Background] Nystrom E, Sjostrom M, Stenlund H, Samuelsson E. ICIQ symptom and quality of life instruments measure clinically relevant improvements in women with stress urinary incontinence. Neurourol Urodyn. 2015 Nov;34(8):747-51. doi: 10.1002/nau.22657. Epub 2014 Aug 22. PMID 25154378